CLINICAL TRIAL: NCT02919098
Title: In-School Evaluation of Bystander: A Game-Based Intervention for Sexual Violence Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB15-1404
Record Dates: First submitted 2016-09-28; First posted 2016-09-29 (Estimated); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Bystander Behavioral Intentions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Two schools (all students grades 9-12) will serve as the intervention group.Participants will complete a baseline survey that will take no longer than 30 minutes. Afterwards, a trained facilitator will delivery a game-based bystander intervention program aimed at teaching students the knowledge and skills to prevent or intervene in instances in sexual harassment and violence among peers. This will last for 4 class periods (approximately 45 minutes each period, 180 minutes total). Afterwards, participants will complete an immediate post-program survey lasting no more than 30 minutes. Three months later, students will fill out an a follow up survey lasting no more than 30 minutes. School staff and administrators will be interviewed to gather their insights on the program's feasibility and acceptability.
  Interventions: Behavioral: Bystander, a game-based bystander intervention program
- Delayed Control (Placebo Comparator): One school (all students grades 9-12) will serve as a delayed control group. Participants will complete a baseline survey that will take no longer than 30 minutes. Afterwards, a trained facilitator will delivery a game-based health program unrelated to sexual health, sexual violence, sexual harassment, and bystander behaviors. This will last for 4 class periods (approximately 45 minutes each period, 180 minutes total). Afterwards, participants will complete an immediate post-program survey lasting no more than 30 minutes. Three months later, students will fill out an a follow up survey lasting no more than 30 minutes.
  After completing the follow-up survey, this group will follow the same procedures to deliver the bystander program and capture data outlined for the intervention group.
  Interventions: Behavioral: Bystander, a game-based bystander intervention program; Behavioral: Infection City, a game-based program about meningitis

INTERVENTIONS:
Behavioral: Bystander, a game-based bystander intervention program — A game-based, high school age-appropriate program delivered by trained facilitators for sexual violence and harassment intervention
Behavioral: Infection City, a game-based program about meningitis — A game-based, high school age-appropriate program delivered by trained facilitators to teach students about meningitis.
  Arms: Delayed Control

SUMMARY:
The investigators have developed a game-based sexual violence prevention program that uses a bystander intervention approach. This program is called Bystander and was designed for use with high school students in grades 9-12. The goal of this research is to evaluate the efficacy and feasibility of Bystander when implemented in a school setting. The research will capture data on knowledge about sexual violence and harassment, as well as attitudes, self-efficacy, perceived social norms and behavioral intentions around bystander behaviors. This research will consist of a baseline survey, program participation, a immediate post-program survey, and a 3-month follow up survey with youth participants. It will also involve qualitative in-depth interviews with school staff and administration about the program.

DETAILED DESCRIPTION:
Using the investigators' experience in game-based learning, digital media, behavior theory, and adolescent sexual and reproductive health, the investigators have developed a digital game-based sexual violence prevention program-Bystander-to be used with high school students to teach them about prosocial bystander behaviors and decrease acceptance of common rape myths. The goal of this research is to evaluate the efficacy and feasibility of Bystander when implemented in a school setting.

This study will evaluate Bystander, a four-module intervention program. Each module is designed to last one school class period. It includes 20 minutes of individual gameplay through an interactive narrative featuring prosocial bystander behaviors and discussions dispelling rape myths. Each module also includes facilitated class discussion about the topics covered that day.

The research team will conduct a pre/post efficacy and feasibility study that will capture data through a pre-, immediate post-, and 3-month follow up survey on knowledge about sexual violence and harassment, as well as attitudes, self-efficacy, perceived social norms and behavioral intentions around bystander behaviors (all measured at pre-, immediate post- and follow-up time points). It will also capture demographic information and previous bystander behaviors at baseline. It will finally involve qualitative in-depth interviews with school staff and administration about the program.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-19 years
* A student in grades 9-12 at one of three identified study site schools
* Able to speak and read English at a 7th grade level
* Provide informed consent and express willingness to complete the follow-up survey.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 601 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
change in bystander behavioral intention | pre, immediate post, 3 month follow up
  measured via validated 11-item Bystander Attitude Scale-Revised by McMahon et al 2014
change in attitudes towards sexual violence and harassment | pre, immediate post, 3 month follow up
  measured via validated 22-item Modified Illinois Rape Myth Acceptance Scale by McMahon 2011

SECONDARY OUTCOMES:
change in knowledge of sexual harassment and violence | pre, immediate post, 3 month follow up
  measured via validated 7-item Legal Knowledge Scale (Maxwell 2003)
change in knowledge of sexual harassment and violence | pre, immediate post, 3 month follow up
  measured via Knowledge of Sexual Violence and Harassment index (Banyard et al 2005)
change in perceived social norms for bystander behaviors | pre, immediate post, 3 month follow up
  measured via validated Social Norms Scale from Gidycz et al 2011
change in self-efficacy for bystander behaviors | pre, immediate post, 3 month follow up
  measured via validated 14-item Bystander Efficacy Scale by Banyard et al 2004
change in self-efficacy for bystander behaviors | pre, immediate post, 3 month follow up
  measured via validated 10-item MVP Efficacy Scale by Ward 2001
change in decisional balance for bystander behaviors | pre, immediate post, 3 month follow up
  measured via validated 10-item Bystander Decisional Balance Scale by Banyard 2004
change in normative beliefs around sexual violence | pre, immediate post, 3 month follow up
  measured via validated 8-item Reaction to Offensive Language Scale--Comfort Subscale by Loh 2005

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Gilliam, MD, MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicao, Chicago, Illinois, United States

REFERENCES:
- [Background] Maxwell, Christopher D., Amanda L. Robinson, and Lori A. Post.
- [Background] McMahon, Sarah, and G. Lawrence Farmer.
- [Background] McMahon S, Allen CT, Postmus JL, McMahon SM, Peterson NA, Lowe Hoffman M. Measuring bystander attitudes and behavior to prevent sexual violence. J Am Coll Health. 2014;62(1):58-66. doi: 10.1080/07448481.2013.849258. PMID 24313697
- [Background] Gidycz CA, Orchowski LM, Berkowitz AD. Preventing sexual aggression among college men: an evaluation of a social norms and bystander intervention program. Violence Against Women. 2011 Jun;17(6):720-42. doi: 10.1177/1077801211409727. Epub 2011 May 12. PMID 21571742
- [Background] Banyard, Victoria L., Elizabethe G. Plante, and Mary M. Moynihan.
- [Background] Ward CL, Flisher AJ, Zissis C, Muller M, Lombard C. Exposure to violence and its relationship to psychopathology in adolescents. Inj Prev. 2001 Dec;7(4):297-301. doi: 10.1136/ip.7.4.297. PMID 11770655
- [Background] Loh C, Gidycz CA, Lobo TR, Luthra R. A prospective analysis of sexual assault perpetration: risk factors related to perpetrator characteristics. J Interpers Violence. 2005 Oct;20(10):1325-48. doi: 10.1177/0886260505278528. PMID 16162492